CLINICAL TRIAL: NCT05599724
Title: Medical Assistance for Procreation Patient Library Targeting Patients With Idiopathic Infertility or Low Ovarian Reserve Before the Age of 35
Brief Title: PMA-FERTITHEQUE Biocollection
Acronym: FERTITHEQUE
Status: Terminated | Type: Observational
Why Stopped: The study was stopped due to organizational challenges affecting participant enrollment, follow-up, and the handling and routing of study samples.
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0053
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Infertility; Infertility Unexplained
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CASE: Patients who did not carry a pregnancy to term
  Interventions: Other: Biocollection
- CONTROL: patients who carried a pregnancy to term
  Interventions: Other: Biocollection

INTERVENTIONS:
Other: Biocollection — For the FERTITHEQUE, will be collected:
  * Clinical characteristics
  * Biological characteristics measured as part of the usual follow-up
  * consultation n°2 : DNA
  * consultation n°2 : plasma
  * consultation n°2 : serum
  * consultation n°2 : vaginal microbiota
  * consultation n°3 : follicular fluid (puncture fluid)
  * consultation n°4 : plasma
  * consultation n°4 : vaginal microbiota.

SUMMARY:
Creation of a patient library in Medically Assisted Procreation to allow the implementation of further research with the following objectives:

* To identify new relevant biomarkers in patients who will carry a pregnancy to term
* To better specify or identify new infertility risk factors
* To identify new relevant biomarkers in patients with reduced ovarian reserve

Four consultations are planned with biological et clinical collection.

DETAILED DESCRIPTION:
* A first initial consultation for prescription of the infertility assessment,
* a consultation 2 summarizing the examinations and delivery of prescriptions
* a blood sample: basal hormonal assessment with AMH (Anti-Mullerian Hormone),
* a urine sample to look for an infection with Chlamydia Trachomatis, which is one of the bacteria responsible for gynecological infections compromising ART.
* an HPV (Human Papillomavirus) test on vaginal swab
* a consultation 3 corresponding to the start of a treatment cycle for IVF with oocyte retrieval at the end of this treatment cycle.
* A consultation lasting 4 to 4-6 weeks to take stock of the success or failure of the ART.
* A pregnancy follow-up consultation if successful, for a pelvic ultrasound, then monthly pregnancy follow-up (one consultation per month).
* As part of the usual ART monitoring, clinical and paraclinical data are collected using the MEDIFIRST software.
* During the inclusion visit, questionnaire => will be completed over an additional time to the consultation if inclusion is desired, inclusion time provided by one of the doctors participating in the study.

For the FERTITHEQUE, will be collected:

* clinical characteristics collected at each consultation as part of the usual follow-up.
* biological characteristics measured as part of the usual follow-up.
* During consultation 2, during a blood test carried out as part of your usual care, additional tubes will be taken (4 to 5 tubes of 10mL) to carry out the banking of DNA (support of genetic information), plasma (plasma library), serum (serotheque).
* During consultation 2, a swab will also be taken from the vaginal microbiota.
* During consultation 3, a conservation of the follicular fluid (puncture fluid) will be carried out.
* During consultation 4, a plasma library will be performed again, whether there is pregnancy or not, as well as a new swab sample for the vaginal microbiota.

Then, as described above, patients are after inclusion as part of the usual IVF follow-up reviewed at 1 month for oocyte retrieval then at 2 months for the follow-up visit allowing observation of success or failure of the treatment cycle.

* If pregnancy is achieved, patients are seen monthly as part of their usual follow-up until delivery.
* If a pregnancy is not achieved, follow-up stops.
* Whether or not a pregnancy is obtained, during the visit at 2 months (V4), a plasma library and a vaginal microbiota are again performed.

ELIGIBILITY:
Inclusion Criteria:

* Signed consent
* Aged 18 to 43
* Infertility for at least 12 months
* Oriented in IVF
* Infertility of unexplained origin or presenting a low ovarian reserve before the age of 35 (AMH<1.1ng and/or CFA<7).

Exclusion Criteria:

* Minor patients or > 43 years old
* Patients under guardianship, curatorship (legal protection)
* Refusal to participate
* Patient unable to consent

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Patients who consented to participate in the study, aged 18 to 43 consulting for infertility of at least 12 months, directed to IVF, of unexplained origin or presenting a low ovarian reserve before 35 years of age (AMH<1.1ng and /or CFA<7).
Sampling Method: Non-Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2022-11-11 (Actual); Primary Completion 2023-04-24 (Actual); Study Completion 2023-04-24 (Actual)

PRIMARY OUTCOMES:
clinical-biological markers | 9 months
  Identify relevant clinical-biological markers (known or not yet known at the time of the constitution of the patient library) allowing to identify the patients who will or will not present a pregnancy at the end of the In Vitro Fertilization treatments

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available after the publication of result and ending fifteen years following the last visit of the last patient
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement